CLINICAL TRIAL: NCT01862393
Title: The Influence of Stimulus Phase Duration on Discomfort and Electrically Induced Torque of Quadriceps Femoris
Brief Title: Stimulus Phase Duration on Discomfort and Electrically Induced Torque of Quadriceps Femoris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Richard Eloin Liebano, Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CAAE - 0081.0.186.000-07
Record Dates: First submitted 2013-05-17; First posted 2013-05-24 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Torque; Pain Perception
Keywords: electrical stimulation; torque

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 400 microseconds (Experimental): Electrically-induced torque generated with stimulus phase duration set at 400 microseconds.
  Interventions: Device: 400 microseconds
- 700 microseconds (Experimental): Electrically-induced torque generated with stimulus phase duration set at 700 microseconds.
  Interventions: Device: 700 microseconds
- 1000 microseconds (Experimental): Electrically-induced torque generated with stimulus phase duration set at 1000 microseconds.
  Interventions: Device: 1000 microseconds

INTERVENTIONS:
Device: 400 microseconds — Neuromuscular electrical stimulation with stimulus phase duration of 400 microseconds
  Arms: 400 microseconds
Device: 700 microseconds — Neuromuscular electrical stimulation with stimulus phase duration of 700 microseconds
  Arms: 700 microseconds
Device: 1000 microseconds — Neuromuscular electrical stimulation with stimulus phase duration of 1000 microseconds
  Arms: 1000 microseconds

SUMMARY:
This study aims to examine the variation in muscle torque and discomfort produced when electrically stimulating quadriceps femoris using pulsed current with three different phase durations in order to establish whether there are any advantages or disadvantages in varying the phase duration over the range examined.

ELIGIBILITY:
Inclusion Criteria:

* sedentary healthy university students.

Exclusion Criteria:

* history of knee surgery or injury,
* musculoskeletal, cardiovascular or neurological disease including impaired sensation.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Torque | During 4 seconds of electrical stimulation
  Torque will be measured using an isokinetic dynamometer. Torque will be registered in Newton meter [N.m]

SECONDARY OUTCOMES:
Discomfort | During 6 seconds of electrical stimulation
  Discomfort will be measured using a 10 cm visual analogue scale (VAS) ranging from zero (no discomfort) to 10 (worst discomfort imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Liebano, PhD, Principal Investigator — Universidade Cidade de Sao Paulo
Locations (1):
- Universidade Cidade de São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided